CLINICAL TRIAL: NCT06240728
Title: A Phase 1a/1b Dose Escalation and Dose Expansion Study of NPX887 in Participants With Solid Tumor Malignancies Known to Express B7-H7/HHLA2
Brief Title: A Study of NPX887 for Participants With Solid Tumors Known to Express B7-H7/HHLA2
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: NextPoint Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NPX887-001
Record Dates: First submitted 2024-01-26; First posted 2024-02-05 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Metastatic Malignant Neoplasm
Keywords: B7-H7; HHLA2; solid tumor malignancies; monoclonal antibody; Dose escalation; Dose expansion; RECIST
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Intervention Model Description: Dose escalation and dose expansion
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- NPX887 Treatment (Experimental): Participants will receive NPX887 by IV infusion every 3 weeks.
  Interventions: Drug: NPX887

INTERVENTIONS:
Drug: NPX887 — NPX887 will be administered by IV infusion every 3 weeks until documented disease progression or participant withdrawal for up to 2 years

SUMMARY:
NPX887 is a human, antagonistic immunoglobulin G1 (IgG1) monoclonal antibody targeting B7-H7 (HHLA2) that may potentiate an anti-tumor immune response. The goal of this first-in-human study is to learn whether NPX887 is safe and tolerable and shows a preliminary efficacy in participants with B7-H7 (HHLA2) expressing tumors at selected dose(s). The main questions it aims to answer are:

* what is an appropriate dose to be given to participants?
* are the side effects of treatment manageable?
* what is the preliminary anti-tumor activities?

Participants who are treated will receive an intravenous (IV) infusion of NPX887 if their disease has not progressed, and be closely monitored by the treating physicians.

DETAILED DESCRIPTION:
This study is comprised of Phase 1a (Dose Escalation) and Phase 1b including Part 1b (Dose Expansion) and Part 1c (Randomized Dose Comparison). Phase 1a will test different doses of NPX887 to determine the optimal dose(s) to continue with in Phase 1b. In the Phase 1b, more participants will be tested to evaluate preliminary activities in multiple disease-specific cohorts and compare the efficacy of the higher and lower doses chosen in Phase 1a.

Throughout the study, safety and preliminary efficacy data will be collected to characterize the clinical activity of NPX887. Samples of blood will be taken to help in an understanding of how NPX887 behaves in the body by assessing the amount of drug in the blood over time, and changes in blood components. Tumor tissue samples will be collected at screening and on-treatment stages for biomarker analysis and pharmacodynamics (PD) evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed recurrent, metastatic solid tumor refractory to, or intolerant of, standard of care therapy in one of the following indications:

  * Phase 1a (Dose Escalation): Non-small cell lung carcinoma (NSCLC), small cell lung carcinoma (SCLC), renal cell carcinoma (RCC), colorectal carcinoma (CRC), gastric and gastro-esophageal carcinoma, esophageal adenocarcinoma, biliary tract cancers, ovarian carcinoma, and other solid tumor types known to express B7-H7/HHLA2.
  * Phase 1b including Part 1b (Dose Expansion) and Part 1c (Randomized Dose Comparison): participants who have clear cell RCC, EGFR mutant lung adenocarcinoma, or gastric/GEJ adenocarcinoma.
  * In Phase 1b, participants must have confirmed B7-H7/HHLA2 expression in their tumor determined via archival tissue IHC testing through a central lab (pre-screening).
* Phase 1a: Evaluable disease (measurable or non-measurable) by RECIST v.1.1 criteria; Phase 1b: Measurable disease by RECIST v1.1 criteria with additional disease-specific enrollment criteria applied to clear cell RCC, EGFR mutant lung adenocarcinoma, or gastric/GEJ adenocarcinoma.
* Eastern Cooperative Oncology Group (ECOG) performance status 0, 1, or 2.
* Ability to understand and the willingness to sign a written informed consent document
* Willing to use highly effective contraceptive measures throughout the trial.

Exclusion Criteria:

* Treatment with any of the following:

  * Systemic anticancer treatment ≤14 days or within 5 half-lives prior to the first dose of study drug, whichever is shorter.
  * Limited-field radiotherapy ≤7 days or extended-field thoracic radiotherapy ≤8 weeks of the first dose of study drug.
* Have any unresolved toxicity of ≥Grade 2 from previous anti-cancer treatment, except for alopecia, chronic stable neuropathy for >4 months, changes in skin pigmentation, or requiring replacement therapy for endocrine abnormalities.
* Participants with known brain metastases are excluded unless they are clinically stable, with no new or enlarging brain metastases as evidenced on MRI during screening.
* History of Grade 3 immune-related pneumonitis or colitis.
* Participants who discontinued prior immunotherapy due to immune-related toxicities, or history of unresolved prior immune-related toxicity except for endocrine abnormalities requiring replacement therapy or vitiligo.
* Known autoimmune disease requiring immunosuppressive treatment requiring the equivalent of more than 10 mg prednisone daily.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2024-01-22 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicity (DLT) | From first dose through 21 days
  Number of participants with DLT in Ph1a
Incidence of treatment-emergent adverse events (AEs) | From first dose up to 24 months
  Number and type of AEs categorized by Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 in Ph1a
Incidence of discontinuations, dosing interruptions, and dose reductions | From first dose up to 24 months
  Number of participants with changes to their dosing schedule as a result of treatment-related AEs in Ph1a
Objective response rate (ORR) | Up to 2 years or until progressive disease, unacceptable toxicity, participant withdraw consent or investigator's decision, whichever occurs first.
  The proportion of participants with best overall response of complete response (CR) or partial response (PR) per RECIST 1.1 in Ph1b
Duration of response (DOR) | Up to 2 years or until progressive disease, unacceptable toxicity, participant withdraw consent or investigator's decision, whichever occurs first.
  The time interval from first occurrence of a documented objective response to the time of disease progression as determined by the Investigator using RECIST 1.1 or death from any cause, whichever comes first, in Ph1b
Disease control rate (DCR) | Up to 2 years or until progressive disease, unacceptable toxicity, participant withdraw consent or investigator's decision, whichever occurs first.
  The proportion of participants with a best ORR + Stable Disease (SD) in Ph1b
Progression-free Survival (PFS) | Up to 2 years or until progressive disease, death, unacceptable toxicity, participant withdraw consent or investigator's decision, whichever occurs first.
  The duration from the start of treatment until tumor progression or death of any cause in Ph1b

SECONDARY OUTCOMES:
Area under the concentration curve (AUC0-24) of NPX887 | Following dosing on day 1 of each 21-day treatment cycles up to Cycle 7, then on day 1 every 3 cycles, up to end of treatment and 90-day follow-up
  Measurement of plasma concentration over time for exposure to NPX887
Maximum plasma concentration (Cmax) of NPX887 | Following dosing on day 1 of each 21-day treatment cycles up to Cycle 7, then on day 1 every 3 cycles, up to end of treatment and 90-day follow-up
  Measurement of plasma concentration over time for exposure to NPX887
Half-life in blood circulation (T1/2) of NPX887 | Following dosing on day 1 of each 21-day treatment cycles up to Cycle 7, then on day 1 every 3 cycles, up to end of treatment and 90-day follow-up
  Measurement of the clearance of NPX887 from plasma over time
Immunogenicity of NPX887 | Following dosing on day 1 of each 21-day treatment cycles up to Cycle 4, then on day 1 every 3 cycles, up to 90-day follow-up
  Number of participants with anti-drug antibodies (ADA)
Overall survival (OS) | From first dose until death from any cause through 24 months
  Average length of survival for treated participants
Incidence of AEs, DLTs, PD changes within the tumor and in blood | From first dose through 21 days, or up to 24 months
  Number of participants with AEs and type, DLTs, and PD changes in Ph1a
ORR, DOR, DCR, and PFS | Up to 2 years or until progressive disease, death, unacceptable toxicity, participant withdraw consent or investigator's decision, whichever occurs first.
  ORR, DOR, DCR, and PFS occur in Ph1a

CONTACTS AND LOCATIONS:
Overall Officials: Leena Gandhi, MD, PhD, Study Director — NextPoint
Locations (8):
- United States (6):
  - Johns Hopkins University Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center (BIDMC), Boston, Massachusetts
  - Albert Einstein Medical College Montefiore Medical Center, The Bronx, New York
  - MD Anderson Cancer Center, Houston, Texas
  - Next Oncology, San Antonio, Texas
  - NEXT Oncology-Fairfax, Fairfax, Virginia
- South Korea (2):
  - Severance Hospital, Yonsei University Health System, Seoul
  - Samsung Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: No